CLINICAL TRIAL: NCT06246149
Title: Adjuvant Tebentafusp (IMCgp100) Versus Observation in HLA-A*02:01 Positive Patients Following Definitive Treatment of High-risk Uveal Melanoma: an EORTC Randomized Phase III Study (ATOM Trial)
Brief Title: Adjuvant Tebentafusp in High Risk Ocular Melanoma
Acronym: ATOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Northwell Health (Other); Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2022-MG; EU trial number (Other: 2023-510333-28-00)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Uveal Melanoma
Keywords: Tebentafusp; Adjuvant setting; Randomized phase III study; non-metastatic uveal melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tebentafusp (Experimental): Participants will receive tebentafusp 20 mcg on week 1, 30 mcg on week 2, 68 mcg on week 3, and 68 mcg weekly thereafter for 6 months i.e., maximum 26 infusions.
  Interventions: Drug: Tebentafusp
- Observation (No Intervention)

INTERVENTIONS:
Drug: Tebentafusp — Tebentafusp will be administered weekly i.v.
  Arms: Tebentafusp

SUMMARY:
At least 50% of patients with high-risk primary uveal melanoma will develop a recurrence following treatment of the primary tumour. Observation is currently the standard of care in the non-metastatic setting. Tebentafusp is the first agent proven to improve overall survival in patients with metastatic uveal melanoma in a randomized trial. Based on the results in the advanced setting, it is hypothesized that treatment with tebentafusp may reduce the risk of development of disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Primary non-metastatic UM, except iris melanoma, after definitive treatment either by surgery or radiotherapy
* Time from primary treatment smaller than 11 weeks (note that the maximum time between primary treatment and randomization is 12 weeks )
* High-risk according to either 1) clinical criteria: TNM (AJCC8) stage III or 2) genetic criteria: monosomy 3 or GEP class 2. Prior to enrolment of the first patient, each site will declare which of the two genetic criteria it uses. Patients with stage I and stage II are only eligible if they meet the genetic criterion declared by the site.
* ECOG performance status of 0 or 1
* 18 years or older
* HLA-A*02:01 positivity by local assessment
* No evidence of UM recurrence, as evidenced by the required baseline imaging performed within 4 weeks prior to randomization
* Adequate organ function
* Time-interval between the end of primary treatment and the randomization less than or equal to 12 weeks
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for women of childbearing potential (WOCBP) within 3 days prior to randomization.
* For patients of childbearing / reproductive potential, agreement to use adequate birth control measures during the study treatment period and for at least 6 months after the last dose of treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.
* For female subjects who are breast feeding, agreement to discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Written informed consent according to ICH/GCP and local regulations

Exclusion Criteria:

* Clinically significant cardiac disease or impaired cardiac function, including any of the following:
* Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade ≥ 2), uncontrolled hypertension, or clinically significant arrhythmia currently requiring medical treatment
* QTcF > 470 msec on screening electrocardiogram (ECG) or congenital long QT syndrome based on at least 3 ECGs obtained over a brief time interval (i.e., within 30 minutes)
* Acute myocardial infarction or unstable angina pectoris < 6 months prior to screening
* Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to randomization
* Any evidence of severe or uncontrolled systemic disease or active infection including hepatitis B, hepatitis C and known active human immunodeficiency virus (HIV) defined as >200 copies of HIV per ml of blood, active bleeding diatheses or renal transplant. NOTE: testing for HIV, HBV, and HCV status prior to enrolment is not necessary unless clinically indicated.
* Participant with history of HBV infection will be eligible if on stable anti-viral therapy for > 4 weeks prior to the planned first dose of study intervention and viral load confirmed as undetectable during Screening.
* Participant with history of HBC infection will be eligible the participant has received curative treatment and viral load was confirmed as undetectable during Screening.
* History of another primary malignancy except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and with the following exception. Patients with a history of another primary cancer treated with curative intent more than 3 years before study entry, who are not receiving any anti-cancer therapy, have a risk of disease recurrence lower than 10% as evaluated by the local Investigator, and who have no toxicity from previous treatment are eligible.
* Participants with active autoimmune disease requiring immunosuppressive treatment, including inflammatory bowel disease (ulcerative colitis or Crohn's disease), within 2 years of screening. NOTE: The following exceptions are permitted:
* Vitiligo
* Alopecia
* Managed hypothyroidism (on stable replacement doses)
* Asymptomatic adrenal insufficiency (on stable replacement doses)
* Psoriasis
* Resolved childhood asthma/atopy
* Well-controlled asthma
* Type I diabetes mellitus
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the trial.
* Known contraindication to imaging tracer or any product of contrast media and MRI and/or CT contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free survival (RFS) | 8.1 years from first patient in
  RFS is defined as the time between randomization and local recurrence, distant recurrence, or death, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | 8.1 years from first patient in
  OS is defined as the time between randomization and death
Occurrence of Adverse Events | 8.1 years from first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting
Health-related Quality of Life | 8.1 years from first patient in
  It will be evaluated using self-administered EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nathan, Principal Investigator — Mount Vernon Cancer Centre, Northwood, UK; Richard D. Carvajal, Principal Investigator — Northwell Health Cancer Institute, NY, USA; Serge Leyvraz, Principal Investigator — Charité Hospital, Berlin, Germany
Locations (13):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (2):
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Hôpital de Paris, Paris
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaets Krankenhaus Eppendorf - Universitaetsklinikum Hamburg-Eppendorf KE - University Cancer Center, Hamburg
  - Universitaetsklinikum Heidelberg - Frauenklinik / Hautklinik, Heidelberg
- Leiden University Medical Centre, Leiden, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Centre - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland
- Spain (2):
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), L'Hospitalet de Llobregat
  - Hospital Clinico Universitario De Valladolid, Valladolid
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- United Kingdom (2):
  - The Clatterbridge cancer Center NHS foundation Trust - Clatterbridge Cancer Center - Liverpool, Liverpool
  - East and North Hertfordshire NHS Trust - Mount Vernon Hospital, Northwood